CLINICAL TRIAL: NCT03149276
Title: Limited English Proficiency Occupational Therapy Patients Receiving Interpreter Services Perception of Quality of Care
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Eileen Turgeon, Occupational Therapist, Rush University Medical Center
Other Study IDs: 14110802-IRB01
Record Dates: First submitted 2017-05-01; First posted 2017-05-11 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Communication Barriers; Occupational Therapy
MeSH Terms: interventions — Occupational Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Limited English Proficiency Group: LEP persons were identified by asking, "What language would you like to receive medical information and services in?" Patients were considered limited English proficient when a non-English language was preferred. Interventions included professional interpreter services and occupational therapy.
  Interventions: Other: Interpreter services
- English Speaking Group: English speaking persons were identified by asking, "What language would you like to receive medical information and services in?" Patients were considered English speaking when the English language was preferred. Intervention included occupational therapy.

INTERVENTIONS:
Other: Interpreter services
  Other Names: Occupational Therapy
  Groups: Limited English Proficiency Group

SUMMARY:
A systematic literature review from March through June 2014 supports the premise that limited English proficiency (LEP) persons face barriers and disparities to medical care that English-speaking persons do not face. Language barriers have a negative impact on health and health care, including lower health status, lower likelihood of having a primary care provider, lower rate of preventative care, higher use rate of diagnostic tests, higher rate of severe psychopathology diagnoses, and higher risk of drug complications . Additionally, LEP persons experience problems with effective communication with providers, inappropriate diagnoses and treatments, lower comprehension of medication instructions and adherence to regimens, fewer follow up visits, low quality care, poorer health outcomes, and low patient satisfaction.

Research has proven a relationship between LEP and health care outcomes, specifically a relationship between positive outcomes and use of professional interpreters. Not sharing a common language creates a barrier to providing safe, effective, client-centered Occupational Therapy (OT) and knowledge of outcome satisfaction for this population. Using trained interpreters would reduce the barriers created by language discordance.

This evidence-based project intends to measures the influence of interpreter service on LEP patients' perceived quality of care using a satisfaction survey. Gathered data will be used to consider development and implementation of practice guidelines for use of professional interpreter services for LEP patients receiving OT services at Midwest Orthopaedics at Rush. Development and implementation of practice guidelines that include use of trained interpreters when providing OT services to LEP patients will facilitate a client-centered approach and improve quality of care for this population.

The project is also being implemented as part of a degree requirement for the Doctorate of Occupational Therapy Program at Chatham University.

DETAILED DESCRIPTION:
The sampling frame will consist of adults, age 18 or older, with limited English proficiency (LEP), with an upper extremity injury or disorder, that have been referred to occupational therapy (OT) at Midwest Orthopaedics at Rush (MOR), require services that span four weeks or more, agree to use of interpreter services, agree to completing a paper and pencil survey at the end of four weeks, and agree to be interviewed after four weeks of occupational therapy services, following completion of the survey. LEP is determined by a preference to receive medical information in a non-English language. Sampling frame is four participants. The sampling frame will be purposive. As LEP individuals present for OT services they will be recruited for participation. Recruitment could happen simultaneously or in tandem.

The comparison group sampling frame will consist of adults, age 18 or older, proficient in English, with an upper extremity injury or disorder, that have been referred to OT at MOR, and require services that span four weeks or more. English proficiency is determined by use of English as preferred language. Sampling frame is four participants. For each LEP individual recruited, the following English-speaking individual will be asked to participate. When participants in each group are recruited, further recruitment will cease. The total sampling frame will be eight. Enlisting an English proficient individual following recruitment of an LEP individual ensures having equal participation in each group.

A paper and pencil survey will be administered in person at MOR after the initial occupational therapy visit and at the end of four weeks of OT services to the 4 Limited English proficient subjects and 4 English-speaking subjects, for 16 completed surveys. Completion will take place in a private room in the OT department. Subjects will self-select a 4 digit identification code that they will write in at the top of the survey. The sole purpose of the code is to match the pre-OT satisfaction survey with the post-OT satisfaction survey. No personal identification markers will be used on the surveys. Interviews will be conducted with each LEP individual following four weeks of OT services and after completion of the paper survey. No personal identification markers will be placed on the interview form. The interviews will be conducted in person at MOR, in a private room in the OT department. The primary investigator will present the open-ended questions with the assistance of Rush University Medical Center (RUMC) interpreter services. The documented data will be reviewed by the primary investigator for emerging themes that may provide insight and additional information.

ELIGIBILITY:
Inclusion Criteria:

* Must be age 18 or older
* Must have a current prescription for occupational therapy (OT) that requires service for four weeks or more that span the six-week length of the project
* Agree to sign the project informed consent form
* Agree to complete the pre-OT satisfaction survey in its entirety at the conclusion of their OT initial evaluation and the post-4 weeks OT satisfaction survey at the end of four weeks of OT service

Additional inclusion criteria for limited English proficiency (LEP) group:

* Agree to use professional interpreter services
* Agree to an interview at the end of four weeks of OT service

Exclusion Criteria:

* Under 18 years of age
* Does not have a current prescription for occupational therapy (OT) that requires service for four weeks or more that span the six-week length of the project
* Refusal to sign the project informed consent form
* Refusal to complete the pre-OT satisfaction survey in its entirety at the conclusion of their OT initial evaluation and the post-4 weeks OT satisfaction survey at the end of four weeks of OT service
* Refusal of LEP participants to use professional interpreter services
* Refusal of LEP participants to be interviewed at the end of four weeks of OT service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Four limited English proficient persons that require occupational therapy services for four or more weeks and four English-speaking persons that require occupational therapy services, for four or more weeks, to serve as a comparison group
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2015-01-06 (Actual); Primary Completion 2015-04-15 (Actual); Study Completion 2015-04-15 (Actual)

PRIMARY OUTCOMES:
Pre-Occupational Therapy Satisfaction Survey | Baseline
  The pre-Occupational Therapy satisfaction survey was developed for this project by the primary investigator to measure perceived satisfaction. The pre-OT satisfaction survey consists of five demographic items and four items that employ a Likert scale rating method. The total quantitative scoring range for the survey is four to twenty, with a score of four indicating the lowest satisfaction and a score of 20 indicating the highest satisfaction. The paper and pencil survey was completed in person by all participants after the initial OT visit. Survey scores of the LEP group were compared to the English-speaking group. Equal or better scores reflect agreement that LEP OT perceive quality of care and satisfaction equal to English-speaking patients.
Post-4 weeks Occupational Therapy Satisfaction Survey | 4 weeks from baseline
  The Post-4 weeks OT satisfaction survey was developed for this project by the primary investigator to measure perceived satisfaction. The survey consists of five demographic items and four items that employ a Likert scale rating method. The total quantitative scoring range for the survey is 4 to 20, with a score of 4 indicating the lowest satisfaction and a score of 20 indicating the highest satisfaction. The post-4 weeks OT satisfaction survey contains three additional items, using a Likert scale rating method to explore qualitative experiences. Total qualitative scoring range for the survey is 3 to 15, with a score of 3 indicating a low belief in the benefits of OT and a score of 15 indicating a high belief in the benefits of OT. Scores of the LEP group were compared to the English-speaking group. Equal or better scores reflect agreement that LEP OT patients receiving IS perceive quality of care and satisfaction equal to English-speaking patients.
Occupational Therapy Satisfaction Interview | 4 weeks from baseline
  Interviews were conducted by the primary investigator, Eileen Turgeon, assisted by Interpreter Services (IS), with each LEP individual following four weeks of OT services and after completion of the post-4 weeks OT satisfaction survey. The interviews were conducted in person. The interview consisted of seven open-ended questions meant to capture the qualitative experience of the use of Interpreter Services during OT service delivery. The literature supports the use of surveys and interviews to gather feedback on LEP patients' perceived quality of care and satisfaction (González et al., 2010; Green et al., 2005; Lee et al., 2002; Shi et al., 2009; Wilson et al., 2005). The primary investigator presented the open-ended questions with the assistance of IS. The recorded interviews were reviewed by this primary investigator for emerging themes to provide insight and additional information.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen D. Turgeon, OTD, Principal Investigator — Rush University Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Occupational Therapy Association. (2014). Occupational therapy practice framework: Domain & process (3rd ed.) [Supplemental Section]. American Journal of Occupational Therapy, 68(Supl. 1), S1-S48.
- [Background] Zuniga GC, Seol YH, Dadig B, Guion WK, Rice V. Progression in understanding and implementing the cultural and linguistic appropriate services standards: five-year follow-up at an academic center. Health Care Manag (Frederick). 2013 Apr-Jun;32(2):167-72. doi: 10.1097/HCM.0b013e31828ef655. PMID 23629039
- [Background] Wilson E, Chen AH, Grumbach K, Wang F, Fernandez A. Effects of limited English proficiency and physician language on health care comprehension. J Gen Intern Med. 2005 Sep;20(9):800-6. doi: 10.1111/j.1525-1497.2005.0174.x. PMID 16117746
- [Background] Wells, S. (2011). American Occupational Therapy Association advisory opinion for the ethics commission: Cultural competency and ethical practice. Bethesda, MD: American Occupational Therapy Association.
- [Background] Wardin K. A comparison of verbal evaluation of clients with limited English proficiency and English-speaking clients in physical rehabilitation settings. Am J Occup Ther. 1996 Nov-Dec;50(10):816-25. doi: 10.5014/ajot.50.10.816. PMID 8947374
- [Background] U.S. News & World Report. (2015). Top-ranked hospitals for orthopedics. Retrieved from http://health.usnews.com/best-hospitals/rankings/orthopedics/data
- [Background] U.S. Department of Commerce, Economics and Statistics Administration, U.S. Census Bureau. (2013). Language use in the United States: 2011 American community survey report (ACS-22). Retrieved from http://www.census.gov/hhes/socdemo/language/
- [Background] U.S. Census Bureau, 2008-2012 American Community Survey. Retrieved from http://factfinder2.census.gov/faces/nav/jsf/pages/index.xhtml
- [Background] The Kawa Model: Culturally Relevant Occupational Therapy. (2010). Retrieved from: http://individual.utoronto.ca/michaeliwama/index.htm
- [Background] Suarez-Balcazar Y, Rodawoski J, Balcazar F, Taylor-Ritzler T, Portillo N, Barwacz D, Willis C. Perceived levels of cultural competence among occupational therapists. Am J Occup Ther. 2009 Jul-Aug;63(4):498-505. doi: 10.5014/ajot.63.4.498. PMID 19708479
- [Background] Shi L, Lebrun LA, Tsai J. The influence of English proficiency on access to care. Ethn Health. 2009 Dec;14(6):625-42. doi: 10.1080/13557850903248639. PMID 19953393
- [Background] Sentell T, Braun KL. Low health literacy, limited English proficiency, and health status in Asians, Latinos, and other racial/ethnic groups in California. J Health Commun. 2012;17 Suppl 3(Suppl 3):82-99. doi: 10.1080/10810730.2012.712621. PMID 23030563
- [Background] Schier JS, Chan J. Changes in life roles after hand injury. J Hand Ther. 2007 Jan-Mar;20(1):57-68; quiz 69. doi: 10.1197/j.jht.2006.10.005. PMID 17254909
- [Background] McLeod, S. (2008). Likert scale. Retrieved from http://www.simplypsychology.org/likert-scale.html
- [Background] Lion KC, Mangione-Smith R, Martyn M, Hencz P, Fernandez J, Tamura G. Comprehension on family-centered rounds for limited English proficient families. Acad Pediatr. 2013 May-Jun;13(3):236-42. doi: 10.1016/j.acap.2012.12.002. Epub 2013 Mar 13. PMID 23491584
- [Background] Lindsay S, Tetrault S, Desmaris C, King GA, Pierart G. The cultural brokerage work of occupational therapists in providing culturally sensitive care. Can J Occup Ther. 2014 Apr;81(2):114-23. doi: 10.1177/0008417413520441. PMID 25004587
- [Background] Lee LJ, Batal HA, Maselli JH, Kutner JS. Effect of Spanish interpretation method on patient satisfaction in an urban walk-in clinic. J Gen Intern Med. 2002 Aug;17(8):641-5. doi: 10.1046/j.1525-1497.2002.10742.x. PMID 12213146
- [Background] Law, M., & MacDermid, J. (2014). Evidence-Based Rehabilitation: A Guide to Practice, Third Edition. Thorofare, NJ: SLACK Incorporated.
- [Background] Karliner LS, Perez-Stable EJ, Gildengorin G. The language divide. The importance of training in the use of interpreters for outpatient practice. J Gen Intern Med. 2004 Feb;19(2):175-83. doi: 10.1111/j.1525-1497.2004.30268.x. PMID 15009797
- [Background] Karliner LS, Napoles-Springer AM, Schillinger D, Bibbins-Domingo K, Perez-Stable EJ. Identification of limited English proficient patients in clinical care. J Gen Intern Med. 2008 Oct;23(10):1555-60. doi: 10.1007/s11606-008-0693-y. Epub 2008 Jul 10. PMID 18618200
- [Background] Karliner LS, Jacobs EA, Chen AH, Mutha S. Do professional interpreters improve clinical care for patients with limited English proficiency? A systematic review of the literature. Health Serv Res. 2007 Apr;42(2):727-54. doi: 10.1111/j.1475-6773.2006.00629.x. PMID 17362215
- [Background] Jacobs E, Chen AH, Karliner LS, Agger-Gupta N, Mutha S. The need for more research on language barriers in health care: a proposed research agenda. Milbank Q. 2006;84(1):111-33. doi: 10.1111/j.1468-0009.2006.00440.x. PMID 16529570
- [Background] Iwama M. Culture and occupational therapy: meeting the challenge of relevance in a global world. Occup Ther Int. 2007;14(4):183-7. doi: 10.1002/oti.234. No abstract available. PMID 17966112
- [Background] Iwama M. Toward culturally relevant epistemologies in occupational therapy. Am J Occup Ther. 2003 Sep-Oct;57(5):582-8. doi: 10.5014/ajot.57.5.582. No abstract available. PMID 14527123
- [Background] Hyman, I. (2009). Literature review: Costs of not providing interpretation in health care. Access Alliance Publication, LR004, June, 1-15.
- [Background] Gonzalez HM, Vega WA, Tarraf W. Health care quality perceptions among foreign-born Latinos and the importance of speaking the same language. J Am Board Fam Med. 2010 Nov-Dec;23(6):745-52. doi: 10.3122/jabfm.2010.06.090264. PMID 21057070
- [Background] Green AR, Ngo-Metzger Q, Legedza AT, Massagli MP, Phillips RS, Iezzoni LI. Interpreter services, language concordance, and health care quality. Experiences of Asian Americans with limited English proficiency. J Gen Intern Med. 2005 Nov;20(11):1050-6. doi: 10.1111/j.1525-1497.2005.0223.x. PMID 16307633
- [Background] Gray B, Stanley J, Stubbe M, Hilder J. Communication difficulties with limited English proficiency patients: clinician perceptions of clinical risk and patterns of use of interpreters. N Z Med J. 2011 Sep 9;124(1342):23-38. PMID 21963923
- [Background] Fryer C, Mackintosh S, Batchelor F, Hill K, Said C. The effect of limited English proficiency on falls risk and falls prevention after stroke. Age Ageing. 2012 Jan;41(1):104-7. doi: 10.1093/ageing/afr127. Epub 2011 Sep 24. No abstract available. PMID 21948856
- [Background] Flores G. The impact of medical interpreter services on the quality of health care: a systematic review. Med Care Res Rev. 2005 Jun;62(3):255-99. doi: 10.1177/1077558705275416. PMID 15894705
- [Background] Cooper, L., & Powe, N. (2004). Disparities in patient experiences, health care processes, and outcomes: The role of patient-provider racial, ethnic, and language concordance. The Commonwealth Fund. Retrieved from http://www.commonwealthfund.org/publications/fund-reports/2004/jul/disparities-in-patient-experiences--health-care-processes--and-outcomes--the-role-of-patient-provide
- [Background] Chan J, Spencer J. Adaptation to hand injury: an evolving experience. Am J Occup Ther. 2004 Mar-Apr;58(2):128-39. doi: 10.5014/ajot.58.2.128. PMID 15068148
- [Background] Case-Smith J. Outcomes in hand rehabilitation using occupational therapy services. Am J Occup Ther. 2003 Sep-Oct;57(5):499-506. doi: 10.5014/ajot.57.5.499. PMID 14527111
- [Background] Burke JP, Gitlin LN. How do we change practice when we have the evidence? Am J Occup Ther. 2012 Sep-Oct;66(5):e85-8. doi: 10.5014/ajot.2012.004432. PMID 22917134
- [Background] Bramberg EB, Sandman L. Communication through in-person interpreters: a qualitative study of home care providers' and social workers' views. J Clin Nurs. 2013 Jan;22(1-2):159-67. doi: 10.1111/j.1365-2702.2012.04312.x. Epub 2012 Nov 21. PMID 23170919
- [Background] Betancourt JR, Green AR, Carrillo JE, Ananeh-Firempong O 2nd. Defining cultural competence: a practical framework for addressing racial/ethnic disparities in health and health care. Public Health Rep. 2003 Jul-Aug;118(4):293-302. doi: 10.1093/phr/118.4.293. PMID 12815076